CLINICAL TRIAL: NCT00374660
Title: Phase I-II Clinical and Pharmacokinetic Study of Irofulven in Combination With Oxaliplatin in Patients With Advanced Solid Tumors
Brief Title: Study of Irofulven in Combination With Oxaliplatin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IROF-017
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Liver Cancer
Keywords: Irofulven; Oxaliplatin
MeSH Terms: conditions — Liver Neoplasms | interventions — Oxaliplatin; irofulven

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Irofulven

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered in a 2-hour infusion on Days 1 and 15 of a 28-day cycle. The dose levels ranged from 40 to 80 mg/m^2 by dose escalations in 10 mg/m2 increments if no dose-limiting toxicity.
Drug: Irofulven — Thirty minutes after completion of oxaliplatin infusion, irofulven will be administered as a 30-minute infusion on Days 1 and 15 of a 28-day cycle. The dose levels ranged from 0.30 to 0.40 mg/kg if no dose-limiting toxicity.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and to investigate the efficacy, safety and pharmacokinetics of irofulven combined with oxaliplatin in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures and treatment.
2. Malignant solid tumor confirmed by a biopsy sample.
3. Pancreatic, endometrial, gastric, and hepatocellular cancer patients that have exhausted standard treatment options.
4. Measurable disease according to RECIST.
5. 18 years of age or older.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0-1.
7. Life expectancy greater than 3 months.
8. Previous anticancer treatment must be discontinued at least 4 weeks prior to first dose of study treatment (6 weeks for mitomycin C, 8 weeks for bicalutamide).
9. Patients of reproductive age must be using effective contraceptive methods.
10. Negative pregnancy test for patients of reproductive potential.

Exclusion Criteria:

1. Prior therapy with irofulven or oxaliplatin.
2. Patients who have had radiation therapy to more than 30% of the bone marrow prior to entry into the study.
3. Prior chemotherapy with nitrosoureas or high dose carboplatin (AUC > 6), prior mitomycin C cumulative dose greater than or equal to 25 mg/m², prior bone marrow transplant or intensive chemotherapy with stem cell support.
4. Presence of any serious concomitant systemic disorders incompatible with the study (e.g., uncontrolled congestive heart failure, active infection).
5. Any previous history of another malignancy (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study entry, unless the active malignancy can be unmistakably identified by evidence such as recent biopsies or tumor specific markers.
6. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry.
7. Pregnant or lactating patients or any patient with childbearing potential not using adequate contraception.
8. Patients with retinopathy or significant visual impairment not correctable by refractory lens will be enrolled on a case by case basis according to the expected benefit ratio, taking into account the malignant disease and the existence of an objective decreased visual acuity and its degree.

Please note: There are additional criteria that must be met in order to be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Confirmed response rate: Hepatocellular Cancer (HCC) Cohort: Response Evaluation Criteria in Solid Tumors (RECIST) criteria. | Every 8 weeks until progression.
Hormone Refractory Prostate Cancer (HRPC) Cohort: Prostate-Specific Antigen Working Group Recommendations (PSAWGR) and RECIST criteria. | Every 8 weeks until progression.

SECONDARY OUTCOMES:
Efficacy: HRPC Cohort: confirmed response rate according to RECIST; progression-free survival (PFS) for progression according to RECIST; new bone lesions or skeletal events; PFS according to PSA progression; overall survival. | Every 8 weeks until progression.
Efficacy: HCC cohort - PFS (RECIST); overall survival | Every 8 weeks until progression.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Bordeaux
  - Clichy
  - Lyon
  - Nice
  - Paris
  - Poitiers
  - Saint-Cloud